CLINICAL TRIAL: NCT03433898
Title: An Open Label, Phase I Study of BI 754091 Monotherapy and Combination Therapy of BI 754091 and BI 754111 in Asian Patients With Advanced Solid Tumours
Brief Title: This Study Aims to Find a Safe and Effective Dose of BI 754091. The Study Also Aims to Find Safe and Effective Doses of BI 754091 and BI 754111 in Combination. This Study is Done in Asian Patients With Different Types of Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1381-0004
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part I - ezabenlimab 240 mg (Experimental): Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours were administered via intravenous infusion with ezabenlimab 240 milligram (mg) on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
  Interventions: Drug: Ezabenlimab
- Part II - ezabenlimab 240 mg + BI 754111 400 mg (Experimental): Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours were administered via intravenous infusion with ezabenlimab 240 milligram (mg) and BI 754111 400 mg on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Part II - ezabenlimab 240 mg + BI 754111 600 mg (Experimental): Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours were administered via intravenous infusion with ezabenlimab 240 milligram (mg) and BI 754111 600 mg on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Part II - ezabenlimab 240 mg + BI 754111 800 mg (Experimental): Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours were administered via intravenous infusion with ezabenlimab 240 milligram (mg) and BI 754111 800 mg on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort A (Experimental): Patients with gastric/esophagogastric junction cancer, with no prior treatment with anti-Programmed cell death protein-1 (PD-1)/Programmed death ligand-1 (PD-L1) antibody, and who had received at least one line of systemic anticancer treatment, excluding adjuvant therapy, were administered via intravenous infusion with ezabenlimab 240 milligram (mg) and BI 754111 600 mg on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort B (Experimental): Patients with esophageal cancer, with no prior treatment with anti-Programmed cell death protein-1 (PD-1)/Programmed death ligand-1 (PD-L1) antibody, and who had received at least one line of systemic anticancer treatment, excluding adjuvant therapy, were administered via intravenous infusion with ezabenlimab 240 milligram (mg) and BI 754111 600 mg on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort C (Experimental): Patients with hepatocellular cancer, with no prior treatment with anti-Programmed cell death protein-1 (PD-1)/Programmed death ligand-1 (PD-L1) antibody, who received at least one line of systemic anticancer treatment, excluding adjuvant therapy, and whose Child-Pugh score is ≤7, were administered via intravenous infusion with ezabenlimab 240 milligram (mg) and BI 754111 600 mg on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111
- Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort D (Experimental): Patients with gastric/esophagogastric junction cancer, esophageal cancer, or hepatocellular cancer, with a prior treatment with anti-Programmed cell death protein-1 (PD-1)/Programmed death ligand-1 (PD-L1) antibody, were administered via intravenous infusion with ezabenlimab 240 milligram (mg) and BI 754111 600 mg on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
  Interventions: Drug: Ezabenlimab; Drug: BI 754111

INTERVENTIONS:
Drug: Ezabenlimab — Solution for infusion
  Other Names: BI 754091
Drug: BI 754111 — Solution for infusion
  Arms: Part II - ezabenlimab 240 mg + BI 754111 400 mg; Part II - ezabenlimab 240 mg + BI 754111 600 mg; Part II - ezabenlimab 240 mg + BI 754111 800 mg; Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort A; Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort B; Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort C; Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort D

SUMMARY:
The main objectives of the BI 754091 monotherapy dose-finding part (Part I) of the trial are to investigate the following items in advanced solid tumours:

* Safety, tolerability, and pharmacokinetics (PK) of BI 754091 as monotherapy.
* Maximum tolerated dose (MTD) and/or recommended dose (RD) of BI 754091 monotherapy.

The main objectives of the Combination dose-finding part (Part II) of the trial are to investigate the following items in advanced solid tumours:

* Safety, tolerability, and PK of the combination treatment of BI 754091 and BI 754111.
* MTD and/or RD of the combination treatment of BI 754091 and BI 754111.

The main objectives of the expansion part (Part III) of the trial are:

* To further investigate the safety, tolerability, and PK of the RD of BI 754091 and BI 754111 combination in patients with gastric/esophagogastric junction cancer, esophageal cancer, hepatocellular cancer or non-small cell lung cancer (NSCLC)
* To explore the efficacy of the RD of the combination of BI 754091 and BI 754111 in patients with gastric/esophagogastric junction cancer, esophageal cancer, hepatocellular cancer or NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Of full age (according to local legislation) at the time of signing of the informed consent form (ICF)
* Women of childbearing potential (WOCBP)1 with negative serum pregnancy test at screening and men able to father a child, who agree to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information. The requirement of contraception does not apply to women of no childbearing potential but they must have an evidence of such at screening
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Patients with measurable lesions according to RECIST v1.1
* Conditions specific to respective part of the trial:

  * Part I (BI 754091 dose-finding part):

    * Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours (any type)
    * For whom no therapy of proven efficacy exists, or who are not amenable to standard therapies.
    * Previous treatment with an anti-PD-1 mAb is allowed as long as the last administration of the anti PD-1 mAb on the previous treatment is a minimum of 28 days prior to the first BI 754091 treatment.
  * Part II (Combination dose-finding part):

    * Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours (any type)
    * For whom no therapy of proven efficacy exists, or who are not amenable to standard therapies.
    * Previous treatment with an anti-PD-1 mAb is allowed as long as the last administration of the anti PD-1 mAb on the previous treatment is a minimum of 28 days prior to the first BI 754091 treatment.
  * Part III (Expansion part):

    * Cohort A: Patients with gastric/esophagogastric junction cancer, with no prior treatment with anti-PD-1/PD-L1 antibody, and who received at least one line of systemic medical treatment excluding adjuvant therapy
    * Cohort B: Patients with esophageal cancer with no prior treatment with anti-PD-1/PD-L1 antibody, and who received at least one line of systemic medical treatment excluding adjuvant therapy
    * Cohort C: Patients with hepatocellular cancer with no prior treatment with anti-PD-1/PD-L1 antibody, who received at least one line of systemic medical treatment excluding adjuvant therapy, and whose Child-Pugh score is 7 or less
    * Cohort D: Patients with gastric/esophagogastric junction cancer, esophageal cancer, or hepatocellular cancer with a prior treatment with anti-PD-1/PD-L1 antibody
    * Cohort E: First line squamous or non-squamous NSCLC patients:

      * Without EGFR mutations or ALK rearrangements
      * PD-L1 expression level <50%
    * All cohorts: Patients with advanced and/or metastatic disease, with at least 1 tumour lesion amenable to biopsy, and must be medically fit for biopsy at screening as determined by investigator and willing to undergo a biopsy before first treatment (if adequate archival tissue is not available) and, unless clinically contraindicated, after 6 weeks on therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0 to 1 at screening

Exclusion Criteria:

* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to study entry or planned within 12 months after screening, e.g. hip replacement
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Previous treatment with study medications in this trial
* Any investigational or anti-tumour treatment within 4 weeks or 5 half-life periods (whichever is shorter) prior to the initiation of trial treatment
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 neuropathy due to prior platinum-based therapy
* (Part II and III only) Prior treatment with anti-LAG-3 agents
* Patients with lung cancer that have epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) rearrangements, unless disease has progressed following available EGFR or ALK targeted therapy
* Presence of other active invasive cancers other than the one treated in this Trial within 5 years Prior to screening, with the exception of appropriately treated basal or squamous-cell carcinoma of the skin or in situ carcinoma of the uterine cervix, or other local tumours considered cured by local treatment
* Untreated brain metastasis(es) that may be considered active. Patients with previously treated brain metastases may participate provided they are stable (i.e., without evidence of PD by imaging for at least 4 weeks prior to the first dose of trial treatment, and any neurologic symptoms have returned to baseline), and there is no evidence of new or enlarging brain metastases
* Inadequate organ function or bone marrow reserve as demonstrated by the following laboratory values:

  * Absolute neutrophil count <1.5 x 10^9/L (<1500/mm^3)
  * Platelet count <100 x 10^9/L (<100,000/mm^3)
  * Haemoglobin <9.0 g/dL
  * Alanine aminotransferase (ALT) >2.5 times the upper limit of normal (ULN) if no demonstrable liver lesion(s) (primary or metastases) or >5 times ULN in the presence of liver lesion(s)
  * Aspartate aminotransferase (AST) >2.5 times ULN if no demonstrable liver lesion(s) or >5 times ULN in the presence of liver lesion(s)
  * Total bilirubin >1.5 times ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin >3.0 times ULN or direct bilirubin >1.5 times ULN
  * Serum creatinine (measured by enzymatic assay, Isotope dilution mass spectroscopy [IDMS] standardized Jaffe assay, or non-IDMS Jaffe assay) >1.5 times ULN or estimated glomerular filtration rate (eGFR) <30mL/min/1.73m^2 (Chronic Kidney Disease Epidemiology [CKD-EPI] Collaboration equation); confirmation of eGFR is only required when creatinine is >1.5 X ULN
  * International normalized ratio (INR) (only tested if clinically indicated) >1.5 times ULN (if treated with anticoagulants, prolonged INR is acceptable)
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) >470 msec
  * Any clinically important abnormalities (as assessed by the investigator) in rhythm, conduction, or morphology of resting ECGs, e.g., complete left bundle branch block, third degree heart block
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval
  * Patients with an ejection fraction <55% or the lower limit of normal of the institutional standard will be excluded. Only in cases where the Investigator (or the treating physician or both) suspects cardiac disease with negative effect on the EF, will the EF be measured during screening using an appropriate method according to local standards to confirm eligibility (e.g., echocardiogram [ECHO], multi-gated acquisition scan [MUGA]). A historic measurement of EF no older than 6 months prior to first administration of study drug can be accepted provided that there is clinical evidence that the EF value has not worsened since this measurement in the opinion of the Investigator or of the treating physician or both.
* History of pneumonitis within the last 5 years
* History of severe hypersensitivity reactions to other mAbs
* History of severe hypersensitivity reactions to the ingredients of study drug
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of study treatment
* Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy, or asthma well controlled with steroids
* Active infection requiring systemic treatment (antibacterial, antiviral, or antifungal therapy) at start of treatment in this trial
* Known history of human immunodeficiency virus (HIV) infection or laboratory evidence of hepatitis virus infection with positive results of hepatitis B surface (HBs) antigen and/or presence of HBc antibody together with HBV-DNA and/or hepatitis C RNA (HIV and hepatitis test results obtained in routine diagnostics are acceptable if done within 14 days before the informed consent date). However, for patients with hepatocellular cancer in Part III Cohorts C and D, patients with HBV and/or HCV infection are allowed. Hepatocellular cancer patients in Part III Cohorts C and D with HBV infection must be receiving effective antiviral therapy (viral load <100 IU/mL)
* Current or history of interstitial lung disease
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes him/her an unreliable trial patient, unlikely to complete the trial, or unable to comply with the protocol procedures. However, for patients with hepatocellular cancer in Part III Cohorts C and D, past chronic alcohol abuse are allowed
* Women who are pregnant, nursing, or who plan to become pregnant during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Japan (6):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Kanagawa Cancer Center, Kanagawa, Yokohama
  - Saitama Cancer Center, Saitama, Kitaadachi-gun
  - Shizuoka Cancer Center, Shizuoka, Sunto-gun
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (4):
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital(Linkou), Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Zettl M, Wurm M, Schaaf O, Mostbock S, Tirapu I, Apfler I, Lorenz IC, Frego L, Kenny C, Thibodeau M, Oquendo Cifuentes E, Reschke M, Moll J, Kraut N, Vogt A, Sedgwick JD, Waizenegger IC. Combination of two novel blocking antibodies, anti-PD-1 antibody ezabenlimab (BI 754091) and anti-LAG-3 antibody BI 754111, leads to increased immune cell responses. Oncoimmunology. 2022 Jun 16;11(1):2080328. doi: 10.1080/2162402X.2022.2080328. eCollection 2022. PMID 35756842
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a Phase I, open-label, non-randomised trial in patients with advanced solid tumours to investigate safety, tolerability, pharmacokinetics (PK), maximum tolerated dose (MTD) and/or recommended dose (RD) of BI 754091 (ezabenlimab) as monotherapy (part I), safety, tolerability, PK and RD of ezabenlimab and BI 754111 as combination therapy (part II), and to further investigate the safety, tolerability, PK and efficacy of the combination of ezabenlimab and BI 754111 at RD (part III).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Part I - ezabenlimab 240 mg | Part II - ezabenlimab 240 mg + BI 754111 400 mg | Part II - ezabenlimab 240 mg + BI 754111 600 mg | Part II - ezabenlimab 240 mg + BI 754111 800 mg | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort A | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort B | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort C | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort D
Started | 7 | 3 | 3 | 3 | 37 | 37 | 20 | 36
Treated | 6 | 3 | 3 | 3 | 36 | 37 | 20 | 36
Completed (Completed 1 year of treatment) | 0 | 0 | 0 | 1 | 3 | 3 | 0 | 3
Not Completed | 7 | 3 | 3 | 2 | 34 | 34 | 20 | 33
Not completed — Progressive disease | 6 | 3 | 3 | 2 | 30 | 29 | 17 | 30
Not completed — Not treated | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 2
Not completed — Fatal adverse event: Acute kidney injury | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): TS included all patients who were documented to have received at least one dose of ezabenlimab or BI 754111. The TS was used for both efficacy and safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I - Ezabenlimab 240 mg | Part II - Ezabenlimab 240 mg + BI 754111 400 mg | Part II - Ezabenlimab 240 mg + BI 754111 600 mg | Part II - Ezabenlimab 240 mg + BI 754111 800 mg | Part III - Ezabenlimab 240 mg + BI 754111 600 mg, Cohort A | Part III - Ezabenlimab 240 mg + BI 754111 600 mg, Cohort B | Part III - Ezabenlimab 240 mg + BI 754111 600 mg, Cohort C | Part III - Ezabenlimab 240 mg + BI 754111 600 mg, Cohort D | Total
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 36 | 37 | 20 | 36 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (15.2) | 65.0 (6.2) | 59.0 (16.1) | 45.7 (26.3) | 57.2 (14.0) | 62.5 (8.6) | 58.9 (12.9) | 60.5 (10.4) | 59.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 10 | 6 | 2 | 7 | 32
  Male | 4 | 2 | 0 | 2 | 26 | 31 | 18 | 29 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 3 | 3 | 3 | 36 | 37 | 20 | 36 | 144
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 6 | 3 | 3 | 3 | 36 | 37 | 20 | 36 | 144

OUTCOME MEASURES:

1. Primary Outcome: Part I: Maximum Tolerated Dose (MTD) of Ezabenlimab
Description: MTD is defined as the highest dose for a given schedule expected to cause <25% risk of the true dose limiting toxicity (DLT) rate being ≥33% during the MTD evaluation period.
  Haematologic DLTs: any Grade 5 toxicity; neutropenia ≥Grade 4 for >5 days; any duration Febrile neutropenia; grade 4 thrombocytopenia or Grade 3 with bleeding or requiring platelet transfusions (any Grade); unexplained Grade 4 anaemia or requiring blood transfusions (any Grade).
  Non-haematological DLTs: aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >3x Upper limit of normal (ULN) and total bilirubin >2x ULN without cholestasis signs; any duration ≥Grade 4 AST or ALT; any ≥Grade 3 non-haematologic toxicity with exceptions; any Grade 4 or 5 adverse event; any duration any Grade 2 pneumonitis; any Grade 2 uveitis, eye pain, or blurred vision not improving to Grade 1 within 2 weeks or requiring systemic treatment; any ≥Grade 2 toxicity causing inability to administer trial drug on Cycle 2 Day 1.
Time Frame: First cycle of treatment: 3 weeks (21 days) following drug administration.
Population: Maximum tolerated dose set (MTDS) restricted to Part I: included all patients who were documented to have received at least one dose of ezabenlimab in Part I and were not replaced for the MTD determination. Patients who discontinued during the first treatment course for reasons other than a DLT were excluded from the determination of the MTD. The MTDS was used for the primary analyses of DLTs and MTD determination.
Measure: Number; unit: Milligram
Arm/Group | Part I - ezabenlimab 240 mg
Number analyzed (Participants) | 6
Milligram | NA — There was no DLT in Part I of this trial during the first cycle and, therefore, an MTD was not reached within the investigated dose range.

2. Primary Outcome: Part I: Number of Patients Experiencing DLTs During the MTD Evaluation Period (First Cycle of Treatment)
Description: Number of patients experiencing DLTs during the MTD evaluation period (first cycle of treatment) is reported.
Time Frame: First cycle of treatment: 3 weeks (21 days) following drug administration.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - ezabenlimab 240 mg
Number analyzed (Participants) | 6
Participants | 0

3. Primary Outcome: Part II: MTD of the Ezabenlimab Plus BI 754111 Combination Therapy
Description: MTD is defined as the highest dose for a given schedule expected to cause <25% risk of the true DLT rate being ≥33% during the MTD evaluation period.
  Haematologic DLTs: any Grade 5 toxicity; neutropenia ≥Grade 4 for >5 days; any duration Febrile neutropenia; grade 4 thrombocytopenia or Grade 3 with bleeding or requiring platelet transfusions (any Grade); unexplained Grade 4 anaemia or requiring blood transfusions (any Grade).
  Non-haematological DLTs: aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >3x Upper limit of normal (ULN) and total bilirubin >2x ULN without cholestasis signs; any duration ≥Grade 4 AST or ALT; any ≥Grade 3 non-haematologic toxicity with exceptions; any Grade 4 or 5 adverse event; any duration any Grade 2 pneumonitis; any Grade 2 uveitis, eye pain, or blurred vision not improving to Grade 1 within 2 weeks or requiring systemic treatment; any ≥Grade 2 toxicity causing inability to administer trial drugs on Cycle 2 Day 1.
Time Frame: First cycle of treatment: 3 weeks (21 days) following drug administration.
Population: Maximum tolerated dose set (MTDS) restricted to Part II: included all patients who were documented to have received at least one dose of ezabenlimab or BI 754111 in Part II and were not replaced for the MTD determination. Patients who discontinued during the first treatment course for reasons other than a DLT were excluded from the determination of the MTD. The MTDS was used for the primary analyses of DLTs and MTD determination.
Measure: Number; unit: Milligram
Groups:
- Part II - ezabenlimab 240 mg + multiple BI 754111 doses: Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours were administered via intravenous infusion with ezabenlimab 240 milligram (mg) and BI 754111 400 mg OR 600 mg OR 800 mg on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
Arm/Group | Part II - ezabenlimab 240 mg + multiple BI 754111 doses
Number analyzed (Participants) | 9
Milligram | NA — There was no DLT in Part II of this trial during the first cycle and, therefore, an MTD was not reached within the investigated dose range.

4. Primary Outcome: Part II: Number of Patients Experiencing DLTs During the MTD Evaluation Period (First Cycle of Treatment)
Description: Number of patients experiencing DLTs during the MTD evaluation period (first cycle of treatment) is reported.
Time Frame: First cycle of treatment: 3 weeks (21 days) following drug administration.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part II - ezabenlimab 240 mg + BI 754111 400 mg | Part II - ezabenlimab 240 mg + BI 754111 600 mg | Part II - ezabenlimab 240 mg + BI 754111 800 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

5. Primary Outcome: Part III: Number of Patients With Objective Response (OR) - Confirmed Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 as Assessed by the Investigator
Description: Number of patients with objective response (OR) - confirmed complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumours (RECIST) Version 1.1 as assessed by the Investigator, is reported.
  CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of the first administration of trial treatment until the date of the last administration of trial treatment + 30 days (residual effect period): up to 49 months.
Population: Treated set (TS) restricted to Part III: included all Part III patients who were documented to have received at least one dose of ezabenlimab or BI 754111. The TS was used for both efficacy and safety analyses. Patients with a post baseline measurement are reported here.
Measure: Count of Participants; unit: Participants
Arm/Group | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort A | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort B | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort C | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort D
Number analyzed (Participants) | 33 | 35 | 20 | 32
Participants | 4 | 8 | 0 | 2

6. Secondary Outcome: Part III: Duration of Response
Description: The duration of response, defined as the interval from the date of first documented PR or CR according to RECIST Version 1.1 as assessed by the Investigator, to the date of progressive disease (PD) or death, is reported.
  For all patients with an OR, the duration of OR was calculated as follows:
  * for patients with PD or death: duration of response [days] = date of outcome - date of first assessment indicating OR + 1,
  * for patients without PD or death: duration of response (censored) [days] = date of outcome - date of first assessment indicating OR + 1, for patients without disease progression or death.
  Kaplan-Meier estimates were used to calculate median duration of OR.
Time Frame: From the date of objective response until first date that death or PD has been documented, up to 1362 days.
Population: Treated set (TS) restricted to Part III: included all Part III patients who were documented to have received at least one dose of ezabenlimab or BI 754111. The TS was used for both efficacy and safety analyses. Patients who had a confirmed or unconfirmed objective response are reported here.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort A | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort B | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort C | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort D
Number analyzed (Participants) | 5 | 10 | 1 | 2
Days | 478.0 [99.0 to 484.0] | 148.0 [100.0 to NA] — Not enough events to calculate the 75th percentile. | 44.0 [44.0 to 44.0] | 209.0 [126.0 to 292.0]

7. Secondary Outcome: Part III: Number of Patients With Disease Control
Description: Number of patients with disease control is reported. Disease control: CR, PR, or stable disease (SD) according to RECIST Version 1.1 as assessed by the Investigator.
  SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 5
Population: Treated set (TS) restricted to Part III: included all Part III patients who were documented to have received at least one dose of ezabenlimab or BI 754111. The TS was used for both efficacy and safety analyses. Patients who had a post baseline measurement are reported here.
Measure: Count of Participants; unit: Participants
Arm/Group | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort A | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort B | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort C | Part III - ezabenlimab 240 mg + BI 754111 600 mg, cohort D
Number analyzed (Participants) | 33 | 35 | 20 | 32
Participants | 15 | 16 | 9 | 7

8. Secondary Outcome: Part I: Number of Patients With OR: Confirmed CR or PR According to RECIST v1.1 as Assessed by the Investigator
Description: Number of patients with OR: confirmed CR or PR according to RECIST v1.1 as assessed by the Investigator, is reported.
  CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of the first administration of trial treatment until the date of the last administration of trial treatment + 30 days (residual effect period): 180 days.
Population: Treated set (TS) restricted to Part I: included all Part I patients who were documented to have received at least one dose of ezabenlimab or BI 754111. The TS was used for both efficacy and safety analyses. Patients who had a post baseline measurement are reported here.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I - ezabenlimab 240 mg
Number analyzed (Participants) | 6
Participants | 0

9. Secondary Outcome: Part II: Number of Patients With OR: Confirmed CR or PR According to RECIST v1.1 as Assessed by the Investigator
Description: as for outcome 8
Time Frame: From the date of the first administration of trial treatment until the date of the last administration of trial treatment + 30 days (residual effect period): up to 389 days.
Population: Treated set (TS) restricted to Part II: included all Part II patients who were documented to have received at least one dose of ezabenlimab or BI 754111. The TS was used for both efficacy and safety analyses. Patients who had a post baseline measurement are reported here.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II - ezabenlimab 240 mg + BI 754111 400 mg | Part II - ezabenlimab 240 mg + BI 754111 600 mg | Part II - ezabenlimab 240 mg + BI 754111 800 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 1

10. Secondary Outcome: Part I: Maximum Measured Concentration of Ezabenlimab in Plasma (Cmax) in the First Cycle of Treatment
Description: Maximum measured concentration of ezabenlimab in plasma (Cmax) in the first cycle of treatment (21 days following drug administration) is reported.
Time Frame: 5 minutes before drug administration and 1, 1.5, 2, 4, 7, 24, 48, 72, 168, 336 and 504 hours (h) after the start of drug administration in the first cycle of treatment.
Population: Pharmacokinetic (PK) analysis set (PKS) restricted to Part I: included all Part I patients in the TS who provided at least one evaluable observation for at least one pharmacokinetic endpoint and no pharmacokinetic relevant protocol deviation. The PKS was used for statistical pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Part I - ezabenlimab 240 mg
Number analyzed (Participants) | 6
microgram/milliliter | 78.6 (33.7)

11. Secondary Outcome: Part II: Maximum Measured Concentration of Ezabenlimab in Plasma (Cmax) in the First Cycle of Treatment
Description: as for outcome 10
Time Frame: as for outcome 10
Population: Pharmacokinetic (PK) analysis set (PKS) restricted to Part II: included all Part II patients in the TS who provided at least one evaluable observation for at least one pharmacokinetic endpoint and no pharmacokinetic relevant protocol deviation. The PKS was used for statistical pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Part II - ezabenlimab 240 mg + BI 754111 400 mg | Part II - ezabenlimab 240 mg + BI 754111 600 mg | Part II - ezabenlimab 240 mg + BI 754111 800 mg
Number analyzed (Participants) | 3 | 3 | 3
microgram/milliliter | 88.6 (15.8) | 164 (16.5) | 93.3 (9.50)

12. Secondary Outcome: Part II: Maximum Measured Concentration of BI 754111 in Plasma (Cmax) in the First Cycle of Treatment
Description: Maximum measured concentration of BI 754111 in plasma (Cmax) in the first cycle of treatment (21 days following drug administration) is reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Part II - ezabenlimab 240 mg + BI 754111 400 mg | Part II - ezabenlimab 240 mg + BI 754111 600 mg | Part II - ezabenlimab 240 mg + BI 754111 800 mg
Number analyzed (Participants) | 3 | 3 | 3
microgram/milliliter | 127 (11.0) | 256 (23.0) | 252 (6.52)

13. Secondary Outcome: Part I: Area Under the Concentration-time Curve of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504) in the First Cycle of Treatment
Description: Area under the concentration-time curve of ezabenlimab in plasma over the time interval from 0 to 504 hours (AUC0-504) in the first cycle of treatment (21 days following drug administration) is reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter
Arm/Group | Part I - ezabenlimab 240 mg
Number analyzed (Participants) | 6
hour*microgram/milliliter | 15300 (46.8)

14. Secondary Outcome: Part II: Area Under the Concentration-time Curve of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504) in the First Cycle of Treatment
Description: as for outcome 13
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter
Arm/Group | Part II - ezabenlimab 240 mg + BI 754111 400 mg | Part II - ezabenlimab 240 mg + BI 754111 600 mg | Part II - ezabenlimab 240 mg + BI 754111 800 mg
Number analyzed (Participants) | 3 | 3 | 3
hour*microgram/milliliter | 17500 (22.1) | 26400 (12.5) | 18300 (5.18)

15. Secondary Outcome: Part II: Area Under the Concentration-time Curve of BI 754111 in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504) in the First Cycle of Treatment
Description: Area under the concentration-time curve of BI 754111 in plasma over the time interval from 0 to 504 hours (AUC0-504) in the first cycle of treatment (21 days following drug administration) is reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter
Arm/Group | Part II - ezabenlimab 240 mg + BI 754111 400 mg | Part II - ezabenlimab 240 mg + BI 754111 600 mg | Part II - ezabenlimab 240 mg + BI 754111 800 mg
Number analyzed (Participants) | 3 | 3 | 3
hour*microgram/milliliter | 19900 (16.4) | 39400 (32.1) | 44200 (8.29)

ADVERSE EVENTS:
Time Frame: From the date of the first administration of trial treatment until the date of the last administration of trial treatment + 30 days (residual effect period): 180 days (part I), up to 389 days (part II), up to approximately 49 months (part III). All-cause mortality was recorded from the start of treatment until the end of the follow-up period, up to approximately 49 months.
Description: Treated set (TS): TS included all patients who were documented to have received at least one dose of ezabenlimab or BI 754111. The TS was used for both efficacy and safety analyses.
  AEs have been reported based on drug dosage. Therefore, all the AEs emerged in any patient belonging to any cohort of part III, have been reported together.
Groups:
- Part III - ezabenlimab 240 mg + BI 754111 600 mg: This arm combines cohort A (patients with gastric/esophagogastric junction cancer), cohort B (patients with esophageal cancer), cohort C (patients with hepatocellular cancer), and cohort D (patients with gastric/esophagogastric junction cancer, esophageal cancer, or hepatocellular cancer).
  Patients with advanced and/or metastatic disease were administered via intravenous infusion with ezabenlimab 240 milligram (mg) and BI 754111 600 mg on day 1 of each 3-week (21 days) cycle.
  Administration was continued until progressive disease, unacceptable toxicity, other withdrawal criteria, or a maximum treatment duration of 1 year. If the patient was benefiting clinically at 1 year, he/she could continue after a case-by-case review with the sponsor.
Arm/Group | Part I - ezabenlimab 240 mg | Part II - ezabenlimab 240 mg + BI 754111 400 mg | Part II - ezabenlimab 240 mg + BI 754111 600 mg | Part II - ezabenlimab 240 mg + BI 754111 800 mg | Part III - ezabenlimab 240 mg + BI 754111 600 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/3 | 3/129
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/3 | 1/3 | 1/3 | 36/129
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 3/3 | 100/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I - ezabenlimab 240 mg (N=6) | Part II - ezabenlimab 240 mg + BI 754111 400 mg (N=3) | Part II - ezabenlimab 240 mg + BI 754111 600 mg (N=3) | Part II - ezabenlimab 240 mg + BI 754111 800 mg (N=3) | Part III - ezabenlimab 240 mg + BI 754111 600 mg (N=129)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal rupture (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 6
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Systemic candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Scrotal mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Arterial stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I - ezabenlimab 240 mg (N=6) | Part II - ezabenlimab 240 mg + BI 754111 400 mg (N=3) | Part II - ezabenlimab 240 mg + BI 754111 600 mg (N=3) | Part II - ezabenlimab 240 mg + BI 754111 800 mg (N=3) | Part III - ezabenlimab 240 mg + BI 754111 600 mg (N=129)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 18
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 0 | 11
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 7
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 12
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 11
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 12
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 7
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 7
Fatigue (General disorders) | 3 | 0 | 0 | 0 | 13
Pyrexia (General disorders) | 0 | 0 | 2 | 2 | 32
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 13
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 8
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 8
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 13
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 8
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 3 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
A Cohort E in part III, composed of first line non-small cell lung cancer patients, was also originally planned. However, the clinical development of the combination therapy of BI 754111 and ezabenlimab was concluded early according to protocol due to lack of efficacy of BI 754111 before Cohort E was initiated, so no patient was enrolled in the cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT03433898/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT03433898/SAP_001.pdf